CLINICAL TRIAL: NCT04705116
Title: COVID-19 Vaccines International Pregnancy Exposure Registry (C-VIPER)
Brief Title: COVID-19 Vaccines International Pregnancy Exposure Registry
Acronym: C-VIPER
Status: Recruiting | Type: Observational
Sponsor: Pregistry (Industry)
Responsible Party: Sponsor
Other Study IDs: PR004
Record Dates: First submitted 2021-01-01; First posted 2021-01-12 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 21 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Vaccinated pregnant women: Pregnant women who received at least one dose of a COVID-19 vaccine from 30 days prior to the first day of the LMP to end of pregnancy.
  Interventions: Biological: COVID-19 vaccine
- Non-vaccinated pregnant women: Pregnant women who have not received a COVID-19 vaccine during pregnancy.

INTERVENTIONS:
Biological: COVID-19 vaccine — At least one dose of a COVID-19 vaccine.
  Groups: Vaccinated pregnant women

SUMMARY:
The objective of the COVID-19 Vaccines International Pregnancy Exposure Registry (C-VIPER) is to evaluate obstetric, neonatal, and infant outcomes among women vaccinated during pregnancy with a COVID-19 vaccine.

Specifically, the C-VIPER will estimate the risk of obstetric outcomes (spontaneous abortion, antenatal bleeding, gestational diabetes, gestational hypertension, intrauterine growth restriction, postpartum hemorrhage, fetal distress, uterine rupture, placenta previa, chorioamnionitis, Caesarean delivery, COVID-19), neonatal outcomes (major congenital malformations, low birth weight, neonatal death, neonatal encephalopathy, neonatal infections, neonatal acute kidney injury, preterm birth, respiratory distress in the newborn, small for gestational age, stillbirth, COVID-19), and infant outcomes (developmental milestones [motor, cognitive, language, social-emotional, and mental health skills], height, weight, failure to thrive, medical conditions during the first 12 months of life, COVID-19) among pregnant women exposed to single (homologous) or mixed (heterologous) COVID-19 vaccine brand series from 30 days prior to the first day of the last menstrual period to end of pregnancy and their offspring relative to a matched reference group who received no COVID-19 vaccines during pregnancy.

DETAILED DESCRIPTION:
Rationale and background: COVID-19 vaccines will be used in pregnant populations. Scientific evidence regarding their safety for pregnant women and the developing fetus is lacking.

Objective: The objective of the COVID-19 Vaccines International Pregnancy Exposure Registry (C-VIPER) is to estimate the risk of obstetric outcomes (spontaneous abortion, antenatal bleeding, gestational diabetes, gestational hypertension, intrauterine growth restriction, postpartum hemorrhage, fetal distress, uterine rupture, placenta previa, chorioamnionitis, Caesarean delivery, COVID-19), neonatal outcomes (major congenital malformations, low birth weight, neonatal death, neonatal encephalopathy, neonatal infections, neonatal acute kidney injury, preterm birth, respiratory distress in the newborn, small for gestational age, stillbirth, COVID-19), and infant outcomes (developmental milestones [motor, cognitive, language, social-emotional, and mental health skills], height, weight, failure to thrive, medical conditions during the first 12 months of life, COVID-19) among pregnant women exposed to single (homologous) or mixed (heterologous) COVID-19 vaccine brand series from 30 days prior to the first day of the last menstrual period (LMP) to end of pregnancy and their offspring relative to a matched reference group who received no COVID-19 vaccines during pregnancy.

Study design: The C-VIPER is an international, non-interventional, post-marketing cohort study designed to collect prospective safety data among women vaccinated with a COVID-19 vaccine during pregnancy or within 30 days prior to the first day of the LMP.

Population: The study population includes 2 cohorts of pregnant women 18 years of age and older matched by country and gestational age (±2 weeks):

* Cohort 1: pregnant women exposed from 30 days prior to the first day of the LMP to end of pregnancy to at least one dose of a COVID-19 vaccine. These participants are enrolled as part of the C-VIPER.
* Cohort 2: pregnant women unexposed to a COVID-19 vaccine during pregnancy. These participants are enrolled through the Pregistry International Exposure Registry (PIPER) with the same methods as those in Cohort 1. Women vaccinated before 30 days prior to the first day of the LMP are eligible for inclusion.

Registration and participation via a website especially developed for the C-VIPER are voluntary. Eligible women can enroll at any time during pregnancy.

Data collection: Pregnancy data are collected at enrollment, monthly, and at the end of pregnancy. Liveborn infants are followed-up and data are collected at birth and then every three months until 12 months of age. Information is obtained directly from the participant. The C-VIPER collects data on potential confounding factors (such as maternal sociodemographic characteristics, occupation, behaviors, reproductive history, chronic conditions, results of SARS-CoV-2 tests before and during this pregnancy, new COVID-19 vaccinations, use of medications and other vaccinations, and measures of healthcare utilization), and information related to obstetric, neonatal, and infant outcomes. Given the international nature of the C-VIPER, the questionnaires are available in the languages spoken where it is conducted. Participant confidentiality and anonymity are strictly upheld.

Analysis: Exposure to the vaccine during specific etiologically relevant periods is considered when estimating the risk for each outcome (e.g., first trimester for miscarriages and malformations). Relative risks are presented unadjusted and adjusted using propensity scores (PS) to account for imbalances in characteristics between the exposed and the reference groups.

Sample size: At least 200 pregnancies exposed to each branded COVID-19 vaccine during the first trimester and 300 exposed thereafter during pregnancy are projected. For each exposed pregnancy, 2 unexposed pregnancies enrolled in the PIPER will be matched by country and gestational age at enrollment (±2 weeks).

Study Milestones: The total duration of the study will be 5 years. Obstetric, neonatal, and infant outcomes will be assessed on an ongoing basis as data become available. Data on pregnancy, neonatal and infant outcomes will be included in the interim reports as soon as available. The first two years will include, primarily, enrollment of pregnancies; the third and fourth years will involve follow-up of pregnancies and newborns; and, the final year, will be for data analyses and publications. Results on pregnancy and neonatal outcomes, even preliminary, are expected within the first year of the study. Annual and semi-annual interim reports will be submitted to the Scientific Advisory Committee (SAC) for their review and feedback as well as abbreviated quarterly progress reports summarizing cumulative results on key outcomes. A final report will be prepared at the end of the study.

Governance: The C-VIPER is conducted by Pregistry and includes an internal Safety Management Team (SMT) of experienced pharmacovigilance professionals and a dysmorphologist who meet regularly to review individual cases and safety signals. Additionally, the C-VIPER is in consultation with experts from relevant fields, such as maternal-fetal medicine, infectious diseases, epidemiology, and biostatistics from academic institutions, private practice, and/or government agencies. These individuals constitute the SAC and will provide an independent review of the C-VIPER data.

ELIGIBILITY:
Inclusion criteria:

Vaccinated population:

* Pregnant at time of enrollment
* Age ≥18 years at time of enrollment
* Signed the informed consent form and submitted the baseline module "COVID-19 Vaccination During This Pregnancy"
* Received at least one dose of a COVID-19 vaccine during pregnancy or within the 30 days prior to the first day of the LMP
* Resident of a country where a Central Institutional Review Board (IRB) or Ethics Committee provided approval to conduct the study or clearance that approval is not required to conduct the study

Efforts will be made to obtain documentary evidence of COVID-19 vaccination.

Comparison population:

* Pregnant at time of enrollment
* Age ≥18 years at time of enrollment
* Signed the informed consent form and submitted the minimum required data in the initial baseline questionnaire
* Have not received a COVID-19 vaccine during pregnancy or within the 30 days prior to the first day of the LMP
* Resident of a country where a Central IRB or Ethics Committee provided approval to conduct the study or clearance that approval is not required to conduct the study

Exclusion criteria:

* Not pregnant at time of enrollment
* Age <18 years at time of enrollment

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Persons assigned gender female at birth.
Study Population: The target study population consists of pregnant women who are 18 years of age and older. The exposed group (Cohort 1) includes pregnant women who received at least one dose of a COVID-19 vaccine from 30 days prior to the first day of the LMP to end of pregnancy. The reference group (Cohort 2) includes pregnant women who have not received a COVID-19 vaccine during pregnancy. Women vaccinated against COVID-19 before 30 days prior to the first day of the LMP are eligible in the reference group. Both cohorts will be matched by country of residence and gestational age at enrollment (±2 weeks).
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Obstetric outcomes | 1 year
  Number of pregnant women vaccinated against COVID-19 and number of pregnant women not vaccinated against COVID-19 who experience spontaneous abortion, antenatal bleeding, gestational diabetes, gestational hypertension, intrauterine growth restriction, postpartum hemorrhage, fetal distress, uterine rupture, placenta previa, chorioamnionitis, Caesarean delivery, or COVID-19.
Neonatal outcomes | 1 year
  Number of newborns of women vaccinated against COVID-19 and number of newborns of women not vaccinated against COVID-19 during pregnancy who are diagnosed with major congenital malformations, low birth weight, neonatal death, neonatal encephalopathy, neonatal infections, neonatal acute kidney injury, preterm birth, respiratory distress in the newborn, small for gestational age, stillbirth, or COVID-19.
Infant weight | 1 year
  Change in length and weight from birth to 3, 6, 9, and 12 months of age among newborns of women vaccinated against COVID-19 during pregnancy and among newborns of women not vaccinated against COVID-19 during pregnancy.
Infant developmental milestones | 1 year
  Change in developmental milestones from baseline at 6, 9, and 12 months based on the tool Caregiver Reported Early Development Instruments among the offspring of women vaccinated against COVID-19 during pregnancy and among offspring of women not vaccinated against COVID-19 during pregnancy.
Infant COVID-19 diagnosis | 1 year
  Number of newborns of women vaccinated against COVID-19 during pregnancy and number of newborns of women not vaccinated against COVID-19 during pregnancy diagnosed with failure to thrive, medical conditions, or COVID-19 during the first year of life.
Infant height | 1 year
  Change in height from birth to 3, 6, 9, and 12 months of age among newborns of women vaccinated against COVID-19 during pregnancy and among newborns of women not vaccinated against COVID-19 during pregnancy.

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Renz, MD, Principal Investigator — Pregistry
Locations (1):
- Pregistry, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wyszynski DF, Bhattacharya M, Martinez-Perez O, Scialli AR, Tassinari M, Bar-Zeev N, Renz C, Hernandez-Diaz S. The COVID-19 Vaccines International Pregnancy Exposure Registry (C-VIPER): Protocol and Methodological Considerations. Drug Saf. 2023 Mar;46(3):297-308. doi: 10.1007/s40264-022-01271-3. Epub 2023 Jan 22. PMID 36682012
- See also: COVID-19 Vaccines International Pregnancy Exposure Registry (C-VIPER) — https://c-viper.pregistry.com